CLINICAL TRIAL: NCT02177864
Title: Health Benefits and Tolerance of Dietary Fiber Supplements in Children
Brief Title: Fiber Health Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Warren Bishop (Other)
Responsible Party: Sponsor-Investigator, Warren Bishop, MD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201202731
Record Dates: First submitted 2014-06-24; First posted 2014-06-30 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber (Experimental)
  Interventions: Dietary Supplement: Fiber
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (low fiber bar)

INTERVENTIONS:
Dietary Supplement: Fiber
  Arms: Fiber
Other: Placebo (low fiber bar)
  Arms: Placebo

SUMMARY:
The investigators hypothesize that fiber supplementation will provide measurable differences in indices of children's health (fewer complaints of abdominal pain and constipation, lower body mass index) compared to placebo.

DETAILED DESCRIPTION:
This prospective study proposes supplementing children with fiber or placebo for four months. Children in elementary school, ages 5-12, will be randomized to receive fiber supplemented bars vs low-fiber snack bars (placebo).

ELIGIBILITY:
Inclusion Criteria:

-Children bewteen ages of 5-12 years

Exclusion Criteria:

* History of allergy/intolerance to components of the snack bars (e.g. celiac disease)
* History of Hisrchsprungs disease, abdominal surgery to intestine or colon
* Unable to take a fiber bar by mouth

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in stool frequency | 4 months
  Weekly stool frequency will be compared between baseline and study end in each group
Change in stool consistency | 4 months
  Stool consistency (using the Bristol scale) will be compared between baseline and study end in each group

SECONDARY OUTCOMES:
Change in weight | 4 months
  Weight will be measured and compared between baseline and study end in each group
Change in quality of life score | 4 months
  Pediatric Quality of Life Survey (PedsQL) score will compared between baseline and study end in each group

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bishop, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States